CLINICAL TRIAL: NCT02809729
Title: Antibiotic Prophylaxis in Oncological Surgery of Breast: Randomized Clinical Trial
Brief Title: Antibiotic Prophylaxis in Oncological Surgery of Breast
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fabiola Soares Moreira Campos (Other)
Responsible Party: Sponsor-Investigator, Fabiola Soares Moreira Campos, Department of gynecology, Universidade do Vale do Sapucai
Organization: Universidade do Vale do Sapucai (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MPRUBENS PRUDENCIO
Record Dates: First submitted 2016-06-19; First posted 2016-06-22 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Breast Neoplasms; Breast-Conserving Surgery; Wound Infection; Antibiotic Prophylaxis
MeSH Terms: conditions — Breast Neoplasms; Wound Infection | interventions — Cefazolin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): The patients will receive 0.9% saline for intravenous bottle with 100ml looks identical to the antibiotic at the start of anesthetic induction
  Interventions: Drug: sterile saline; Procedure: oncologic breast surgery; Other: Microbiology
- cefazolin (Active Comparator): The patients will receive 2 g of cefazolin diluted in 0.9% saline by endovenous at the start of anesthetic induction
  Interventions: Drug: Cefazolin; Procedure: oncologic breast surgery; Other: Microbiology

INTERVENTIONS:
Drug: Cefazolin — 2 g of cefazolin diluted in 0.9% saline by endovenous, once, at the moment of anesthetic induction
  Arms: cefazolin
Drug: sterile saline — 0.9% saline sterile by endovenous, once, at the moment of anesthetic induction
  Arms: placebo
Procedure: oncologic breast surgery — The patient will be submitted to a conservative oncologic breast surgery
Other: Microbiology — Samples for quantitative cultures will be obtained in the operating room before antisepsis and the end of surgery. A sample is also collected with the same patterning, on the first postoperative day, immediately after the removal of the dressing placed in the operating room. Will be passed in a standardized manner, a sterile swab soaked in saline over a standard 5cm by 10cm area determined by a field fenestrated sterile filter paper.

SUMMARY:
Breast cancer is the most frequent malignancy in the female population Brazilian, except non-melanoma skin tumors. Surgery plays an important role in regional spot disease control and the definition of parameters for the adjuvant treatment indication. Surgical site infections (SSI) are defined as wound infections occur following invasive procedures, corresponding to 14-16% of all infections nosocomial in hospitalized patients, the most common among patients surgical. SSIs should be examined as potential wound contamination surgical, understood as the number of micro-organisms in the body and / or tissue being operated. Considering this aspect, the cancer surgery breast are classified by their potential for contamination by clean. The use of antibiotics to prevent the SSI in mastectomies is not standardized in Handbook of National Health Surveillance Agency due to the effectiveness of undocumented prophylaxis Thus the use of antibiotics may vary among services. So this randomized clinical trial to evaluate the influence of the use of Prophylactic antibiotics in SSI rates in oncological breast surgery.

DETAILED DESCRIPTION:
KIND OF STUDY:

Primary, clinical, prospective, randomized, two-parallel-group, double-blind, controlled, interventional, analytical. SAMPLE CALCULATION: based on proportions observed in a previous study with and without antibiotic use in breast surgery (VEIGA-Filho, 2010) the number calculated patients per group was 62, with a significance level of 5% and power 80% of the test. SELECTION: will be selected in Mastology outpatient clinics 124 female patients to be undergoing breast surgery for malignancy. The selection of patients will be divided in two groups PLACEBO (N = 62): receive 0.9% saline 100 ml intravenously and CEFAZOLIN GROUP (N = 62): receive 2 g of cefazolin diluted in 0.9% saline by endovenous. In both groups will be passed in a standardized manner, a sterile swab soaked in saline over a standard 5cm by 10cm area determined by a field fenestrated sterile filter paper. Preoperatively will default collection in the region higher interquadrantes breast to be operated immediately above areolopapilar complex, which is not included in the designated area for collection. At end surgery and also in the first postoperative day, the sterile field will be positioned with fenestration on the wound. Tha material will be Standard microbiological methods used to identify microoganismos. 0.2 ml aliquots of each sample are plated on agar media hypertonic mannitol, selective for Staphylococcus sp, Sabouraud agar with chloramphenicol (0.05mg / ml), selective for fungi, agar EMB Teague, selective for enterobacteria, and agar blood, for the presence of hemolytic colonies. After 48 hours, the reading of the number of colony forming units will be held by a microbiologist. Patients are regularly monitored for the occurrence of infection, once a week for the first 30 days by a single surgeon. They will be used and the definitions of surgical site infection classifications adopted by CDC

ELIGIBILITY:
Inclusion Criteria:

* female patients who will undergo breast surgery for cancer evil, between 20 and 75 years, without any restriction as to ethnicity, education or social class;

Exclusion Criteria:

* Patients with BMI greater than 30 kgm 2;
* Patients undergoing neoadjuvant chemotherapy;
* Patients that will undergo immediate breast reconstruction procedures;
* Patients suffering from diabetes mellitus insulin-dependent;
* Patients classified as ASA III or higher
* Patients that postoperative antibiotic therapy have indication by another

clinical complication (cystitis, pneumonia, etc.);

-Patients to withdraw informed consent at any stage of the study;

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2015-01; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
surgical site infection in oncologic breast surgery | up to 30 days
  To evaluate the influence of antibiotic prophylaxis in surgical site infection rates

SECONDARY OUTCOMES:
cutaneous colonization in oncologic breast surgery | intraoperative and the first postoperative day.
  To evaluate the microbiota that infects the skin in oncological breast surgery

CONTACTS AND LOCATIONS:
Overall Officials: FABIOLA SM CAMPOS, MD, Study Chair — department of gynecology and obstetrics
Locations (1):
- Universidade Do Vale Do Sapucai, Pouso Alegre, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No